CLINICAL TRIAL: NCT07067008
Title: Measurement of Intraocular Pressure (With Non-contact Tonometer) in Patients Undergoing Laminectomy in the Prone Position: A Clinical Study
Brief Title: Measurement of Intraocular Pressure in Patients Undergoing Laminectomy in the Prone Position
Status: Not yet recruiting | Type: Observational
Sponsor: Elazıg Fethi Sekin Sehir Hastanesi (Other)
Responsible Party: Sponsor
Other Study IDs: FSCH-SB-2024/07
Record Dates: First submitted 2025-07-04; First posted 2025-07-15 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Laminectomy; Intraocular Pressure; Prone Position
Keywords: Prone Position; Intraocular Pressure; Laminectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 will include those with a BMI of 40 kg/m2 and above.
- Group 2 will include those with a BMI below 40 kg/m2.

SUMMARY:
Laminectomy surgeries, typically performed for lumbar disc herniation and spinal disorders, are often lengthy surgical procedures requiring patients to be in the prone position. While this position provides better visibility of the surgical field, it can lead to physiological changes in intraocular pressure (IOP) in anesthetized patients. An increase in IOP, though rare, has the potential to cause severe ocular complications such as postoperative vision loss (POVL), which is one of the most feared complications after spinal surgery.

One of the main mechanisms of IOP elevation in the prone position is the impediment of venous return in the head and neck region due to gravity, leading to an increase in episcleral venous pressure. Additionally, direct mechanical pressure on the face and globe can also increase IOP. Anesthesia management can also play a role in IOP dynamics by affecting intrathoracic pressure and venous return. This complex interaction necessitates careful monitoring of eye health in anesthetized patients in the prone position. Non-contact tonometers offer a non-invasive, rapid, and reliable method for IOP measurement. They are particularly advantageous for repeated measurements in anesthetized patients. This clinical study aims to evaluate changes in IOP using a non-contact tonometer in patients undergoing laminectomy in the prone position and to identify anesthesia- and patient-related factors influencing these changes. The data obtained will contribute to the development of anesthesia and positioning strategies aimed at reducing the risk of ocular complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for laminectomy surgery under general anesthesia

Patients with ASA physical status I-II-III

Patients who can cooperate postoperatively

Patients without eye diseases or conditions affecting eye physiology (such as glaucoma)

Patients who have not undergone eye surgery

Patients who consent to participate in the study

Exclusion Criteria:

* Patients scheduled for laminectomy surgery but not receiving general anesthesia

Patients with ASA physical status IV-V

Patients who do not consent to participate in the study

Patients who cannot cooperate postoperatively

Patients with eye diseases or conditions affecting eye physiology (such as glaucoma)

Patients who have undergone eye surgery

Patients from whom consent cannot be obtained

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for laminectomy surgery under general anesthesia.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Intraoperative IOP Measurement Schedule After Induction: Intraocular pressure (IOP) is measured non-contact using a tonometer. Intraoperative 1st Hour: After Prone Positioning: | half an hour

IPD SHARING:
Plan to Share IPD: Undecided
Researchers' Interests and Time Constraints

REFERENCES:
- [Background] Kim YS, Seo KH, Jeon YS, In JH, Jung HS, Park YJ, Jun EH, Yu E. Effects of Positive End-Expiratory Pressure on Intraocular Pressure during One-Lung Ventilation in the Lateral Decubitus Position-A Prospective Randomized Trial. Medicina (Kaunas). 2022 Jul 15;58(7):940. doi: 10.3390/medicina58070940. PMID 35888659
- [Background] Saoulidou EN, Giavi VD, Paidakakos NA, Papaconstantinou DS, Dimakopoulou AN, Matsota PK. Effect of Prone Position on Intraocular Pressure in Patients Undergoing Nonocular Surgery: A Systematic Review. Cureus. 2025 May 6;17(5):e83617. doi: 10.7759/cureus.83617. eCollection 2025 May. PMID 40351490